CLINICAL TRIAL: NCT00766675
Title: Ultracet (Tramadol HCL [37.5 mg]/Acetaminophen [325 mg]) Combination Tablets in the Treatment of the Pain of Fibromyalgia
Brief Title: An Efficacy Study of Combination of Tramadol and Acetaminophen Tablets in the Treatment of Participants With Fibromyalgia Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015319; TRAMMAPPAI4033
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Results first posted 2013-07-03 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2013-05

CONDITIONS: Pain; Fibromyalgia
Keywords: Pain; Fibromyalgia; Ultracet; Tramadol Hydrochloride; Acetaminophen
MeSH Terms: conditions — Pain; Fibromyalgia | interventions — Tramadol; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tramadol hydrochloride/acetaminophen (Experimental): Tramadol hydrochloride/acetaminophen oral tablet will be administered as 37.5 /325 milligram respectively once daily for Day 1-3, twice daily for Day 4-6 and thrice daily for Day 7-56.
  Interventions: Drug: Tramadol hydrochloride; Drug: Acetaminophen

INTERVENTIONS:
Drug: Tramadol hydrochloride — Tramadol hydrochloride oral tablet will be administered at a dose of 37.5 milligram as, once daily for Day 1-3, twice daily for Day 4-6 and thrice daily for Day 7-56.
Drug: Acetaminophen — Acetaminophen oral tablet will be administered at a dose of 325 milligram as, once daily for Day 1-3, twice daily for Day 4-6 and thrice daily for Day 7-56.

SUMMARY:
The purpose of this study is to evaluate the analgesic effect of combination of tramadol hydrochloride and acetaminophen in participants for treatment of fibromyalgia pain (chronic widespread pain and presence of tender points).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention) and multi-center (conducted in more than one center) study of combination of tramadol hydrochloride and acetaminophen in treatment of participants with pain of fibromyalgia. The duration of this study will be 56 days per participant. The study consists of 2 parts: Screening (that is, 3 weeks before study commences on Day 1) and Treatment (that is, up to Day 56). All the eligible participants will receive oral tablet for combination of tramadol hydrochloride and acetaminophen. Rescue medication (a medication intended to relieve symptoms immediately) of tylenol (500 milligram, up to 6 oral tablets daily) will be permitted throughout the study duration. Efficacy of the participants will primarily be evaluated by Pain Visual Analog Scale. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the American College of Rheumatology 1990 criteria for the classification of fibromyalgia (that are, Participants must have had widespread pain [pain in three quadrants and in the axial skeleton] for at least three months and pain on digital palpation in 11 or more of the 18 tender-point sites
* Female participants must not be pregnant, breast feeding or postmenopausal for at least one year
* Participant must be able to take oral medication
* Participants must have completed the Screening or wash-out procedures and have a visual analog scale score greater than or equal to 40 milliliter
* Fail to non-opioid analgesics

Exclusion Criteria:

* Participants who previously failed tramadol hydrochloride therapy or those who discontinued tramadol hydrochloride due to adverse events
* Participants diagnosed with either any active connective tissue or musculo-skeletal diseases, or malignancy or history of malignancy within past 5 years, or painful, symptomatic osteoarthritis, or regional periarticular pain syndromes, spondyloarthropathy and major endocrine disease
* Participants who currently have more severe pain than the pain of fibromyalgia
* Participants who have taken antidepressants, cyclobenzaprine or anti-epileptic drugs for pain within three weeks of the Treatment Phase
* Participants who have taken short-acting analgesics, topical medications and anesthetics and/or muscle relaxants for a period of less than 21 days of the given medication prior to the Treatment Phase

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan Ltd Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd

RESULTS

PARTICIPANT FLOW:
Groups:
- Tramadol Hydrochloride/Acetaminophen: Tramadol hydrochloride/acetaminophen oral tablet was administered as 37.5 /325 milligram respectively once daily for Day 1-3, twice daily for Day 4-6 and thrice daily for Day 7-56.
Period: Overall Study
Arm/Group | Tramadol Hydrochloride/Acetaminophen
Started | 80
Completed | 40
Not Completed | 40
Not completed — Adverse Event | 16
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 11
Not completed — Protocol Violation | 8
Not completed — Participant took prohibited medication | 1
Not completed — Receive other anti-neoplastic treatment | 1
Not completed — Insufficient therapy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tramadol Hydrochloride/Acetaminophen
Number analyzed (Participants) | 80
Age Continuous [Mean (Standard Deviation); unit: Years] | 50.4 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 6
Pain Visual Analog Scale at Baseline [Mean (Standard Deviation); unit: Units on a scale] — Assessed by 100 mm of VAS from 0 to 100, where 0 mm=no pain and 10 mm=worse pain.
  Units on a scale | 71.3 (18.22)

OUTCOME MEASURES:

1. Primary Outcome: Pain Visual Analog Scale Score at Day 14
Description: Pain visual analog scale was used to assess the amount of pain recently experienced (within the last 48 hours) by marking a slash through the line of a 100 millimeter (mm) scale measuring pain from "no pain (0 mm)" to "worst possible pain (100 mm)".
Time Frame: Day 14
Population: Intent to treat (ITT) population included all enrolled participants. 'N' (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Millimeter (mm)
Arm/Group | Tramadol Hydrochloride/Acetaminophen
Number analyzed (Participants) | 73
Millimeter (mm) | 53.0 (20.12)

2. Primary Outcome: Pain Visual Analog Scale Score at Day 28
Description: as for outcome 1
Time Frame: Day 28
Population: The ITT population included all enrolled participants. 'N' (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Millimeter (mm)
Arm/Group | Tramadol Hydrochloride/Acetaminophen
Number analyzed (Participants) | 73
Millimeter (mm) | 49.6 (20.95)

3. Primary Outcome: Pain Visual Analog Scale Score at Day 56
Description: as for outcome 1
Time Frame: Day 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Millimeter (mm)
Arm/Group | Tramadol Hydrochloride/Acetaminophen
Number analyzed (Participants) | 73
Millimeter (mm) | 44.9 (20.95)

4. Secondary Outcome: Number of Participants With Categorical Scores on Pain Relief Rating Scale
Description: Pain Relief Rating Scale was used to measure the amount of pain relief experienced (on average) relative to the no-medication Screening or wash-out phase using a 6-point Likert scale ranging from (-) 1 to 4 and rated as (-) 1=worse, 0=None, 1=Slight, 2=moderate,3=a lot and 4=complete.
Time Frame: Day 14, 28 and 56
Population: The ITT population included all enrolled participants.
Measure: Number; unit: Participants
Arm/Group | Tramadol Hydrochloride/Acetaminophen
Number analyzed (Participants) | 80
Participants
  A lot:Day 14 | 12
  Moderate:Day 14 | 19
  Slight:Day 14 | 24
  None:Day 14 | 4
  Worse:Day 14 | 2
  Missing:Day 14 | 19
  A lot:Day 28 | 17
  Moderate:Day 28 | 23
  Slight:Day 28 | 14
  None:Day 28 | 5
  Worse:Day 28 | 3
  Missing:Day 28 | 18
  A lot:Day 56 | 25
  Moderate:Day 56 | 13
  Slight:Day 56 | 18
  None:Day 56 | 9
  Worse:Day 56 | 3
  Missing:Day 56 | 12

5. Secondary Outcome: Tender-Point Evaluation/ Myalgic Score
Description: Eighteen tender-point sites were evaluated by digital palpation for pain by the same Investigator at each site. The Investigator rated the participant's response to digital palpation on a scale from 0 (no pain [participant did not have a tender point]) to 3 (participant withdrawn or flinched). Total myalgic score was the sum of tender-point pain ratings.The total tender-Point score ranges from 0 to 18, and the total myalgic score ranges from 0 to 54. Higher score indicates worsening.
Time Frame: Baseline and Day 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride/Acetaminophen
Number analyzed (Participants) | 51
Units on a scale
  Tender-Point Evaluation (right side):Baseline | 7.9 (1.2)
  Myalgic Score (right side):Baseline | 13.6 (4.0)
  Tender-Point Evaluation (left side):Baseline | 7.8 (1.2)
  Myalgic Score (left side):Baseline | 13.1 (4.1)
  Tender-Point Evaluation (right side):Day 56 | 4.9 (2.5)
  Myalgic Score (right side):Day 56 | 7.0 (5.3)
  Tender-Point Evaluation (left side):Day 56 | 5.1 (2.4)
  Myalgic Score (left side):Day 56 | 7.2 (5.2)

6. Secondary Outcome: Sleep Questionnaire: Number of Hours to Fall Asleep and Participant Slept
Description: The patient assessment sleep questionnaire consisted of 12-Questions (Q) to evaluate the participant's sleep habits out of which Q1 was "How long did it usually take for participant to fall asleep during the past 4 weeks" and Q2 was "On the average, how many hours did participant sleep each night during the past 4 weeks".
Time Frame: Baseline and Day 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Tramadol Hydrochloride/Acetaminophen
Number analyzed (Participants) | 51
Hours
  Question 1: Baseline | 3.2 (1.3)
  Question 2: Baseline | 5.4 (1.5)
  Question 1: Day 56 | 2.2 (1.2)
  Question 2: Day 56 | 6.4 (1.3)

7. Secondary Outcome: Participant Assessment Sleep Questionnaire Score
Description: Sleep questionnaire consisted of 12-Questions (Q), Q3-Q12 were related to "How often during past 4 weeks did participant felt" and are as: Q3: sleep not quiet, Q4: get enough sleep to feel rested upon waking in morning, Q5: awaken short of breath or with headache, Q6: feel drowsy or sleepy, Q7: have trouble falling asleep, Q8: awaken during sleep time and have trouble falling asleep again, Q9: trouble staying awake during day, Q10: snore, Q11: take naps during day, Q12: get amount of sleep needed. Score ranged from 1= all the time to 6 = none of the time, higher score indicates improvement.
Time Frame: Baseline and Day 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride/Acetaminophen
Number analyzed (Participants) | 51
Units on a scale
  Question 3: Baseline | 2.5 (1.3)
  Question 4: Baseline | 4.5 (1.3)
  Question 5: Baseline | 3.8 (1.6)
  Question 6: Baseline | 2.9 (1.5)
  Question 7: Baseline | 2.9 (1.6)
  Question 8: Baseline | 2.9 (1.5)
  Question 9: Baseline | 3.5 (1.6)
  Question 10: Baseline | 3.4 (1.5)
  Question 11: Baseline | 3.3 (1.7)
  Question 12: Baseline | 4.7 (1.3)
  Question 3: Day 56 | 3.8 (1.3)
  Question 4: Day 56 | 3.5 (1.4)
  Question 5: Day 56 | 4.9 (1.1)
  Question 6: Day 56 | 4.3 (1.3)
  Question 7: Day 56 | 4.2 (1.5)
  Question 8: Day 56 | 4.4 (1.3)
  Question 9: Day 56 | 4.4 (1.4)
  Question 10: Day 56 | 4.6 (1.1)
  Question 11: Day 56 | 4.2 (1.4)
  Question 12: Day 56 | 3.8 (1.6)

8. Secondary Outcome: Total Fibromyalgia Impact Questionnaire (FIQ) Score
Description: The FIQ was 19-item questionnaire which measured participant status, progress and outcomes. First 10 items made up of a physical functioning scale, ranging from 0 (always) to 3 (never). Items 11 and 12 asked participants to mark the number of days they felt well (0-7 days) and missed work (0-5 days). Items 13-19 were measured using 10 centimeter (cm) visual analog scale, score ranging from 0 cm (no) to 10 cm (very). Total FIQ score ranged from 0 -100 which was calculated as sum of final scores for item 1-10, 11 and 12, and individual score for item 13-19, and higher score indicates worsening.
Time Frame: Baseline and Day 56
Population: The ITT population included all enrolled participants. 'N' (number of participants analyzed) signifies the participants evaluable for this measure and "n" signifies those participants who were evaluated for this measure at the specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride/Acetaminophen
Number analyzed (Participants) | 73
Units on a scale
  Baseline (n=73) | 6.1 (1.55)
  Day 56 (n=51) | 4.0 (1.94)

9. Secondary Outcome: Number of Participants With Physician Global Assessment
Description: The treating physician rated the participant's condition on Day 1 before the start of treatment and each return visit. The assessment included how the drug controlled the pain (Question 1 [Q1]), adverse event (Question 2 [Q2]), and overall evaluation (Question 3 [Q3]), and participant's condition was indicated as very good, good, moderate, poor and very poor.
Time Frame: Day 14, 28 and 56
Population: The ITT population included all enrolled participants.
Measure: Number; unit: Participants
Arm/Group | Tramadol Hydrochloride/Acetaminophen
Number analyzed (Participants) | 80
Participants
  Q1: Very good (Day 14) | 2
  Q1: Good (Day 14) | 18
  Q1: Moderate (Day 14) | 30
  Q1: Poor (Day 14) | 10
  Q1: Very poor (Day 14) | 2
  Q1: Missing (Day 14) | 18
  Q2: Very good (Day 14) | 19
  Q2: Good (Day 14) | 23
  Q2: Moderate (Day 14) | 14
  Q2: Poor (Day 14) | 4
  Q2: Very poor (Day 14) | 2
  Q2: Missing (Day 14) | 18
  Q3: Very good (Day 14) | 3
  Q3: Good (Day 14) | 14
  Q3: Moderate (Day 14) | 34
  Q3: Poor (Day 14) | 10
  Q3: Very poor (Day 14) | 1
  Q3: Missing (Day 14) | 18
  Q1: Very good (Day 28) | 3
  Q1: Good (Day 28) | 20
  Q1: Moderate (Day 28) | 19
  Q1: Poor (Day 28) | 7
  Q1: Very poor (Day 28) | 0
  Q1: Missing (Day 28) | 31
  Q2: Very good (Day 28) | 14
  Q2: Good (Day 28) | 22
  Q2: Moderate (Day 28) | 11
  Q2: Poor (Day 28) | 2
  Q2: Very poor (Day 28) | 0
  Q2: Missing (Day 28) | 31
  Q3: Very good (Day 28) | 3
  Q3: Good (Day 28) | 23
  Q3: Moderate (Day 28) | 17
  Q3: Poor (Day 28) | 6
  Q3: Very poor (Day 28) | 0
  Q3: Missing (Day 28) | 31
  Q1: Very good (Day 56) | 5
  Q1: Good (Day 56) | 20
  Q1: Moderate (Day 56) | 18
  Q1: Poor (Day 56) | 8
  Q1: Very poor (Day 56) | 1
  Q1: Missing (Day 56) | 28
  Q2: Very good (Day 56) | 13
  Q2: Good (Day 56) | 22
  Q2: Moderate (Day 56) | 13
  Q2: Poor (Day 56) | 2
  Q2: Very poor (Day 56) | 2
  Q2: Missing (Day 56) | 28
  Q3: Very good (Day 56) | 4
  Q3: Good (Day 56) | 26
  Q3: Moderate (Day 56) | 15
  Q3: Poor (Day 56) | 6
  Q3: Very poor (Day 56) | 1
  Q3: Missing (Day 56) | 28

10. Secondary Outcome: Number of Participants With Subject's Global Assessment
Description: Participants indicated their condition on Day 1 before the start of treatment and each return visit. The assessment included how the drug controlled the pain (Question 1 [Q1]), adverse event (Question 2 [Q2]), and overall evaluation (Question 3 [Q3]), and participants indicated their condition as very good, good, moderate, poor and very poor.
Time Frame: Day 14, 28 and 56
Population: The ITT population included all enrolled participants.
Measure: Number; unit: Participants
Arm/Group | Tramadol Hydrochloride/Acetaminophen
Number analyzed (Participants) | 80
Participants
  Q1: Very good (Day 14) | 5
  Q1: Good (Day 14) | 8
  Q1: Moderate (Day 14) | 32
  Q1: Poor (Day 14) | 15
  Q1: Very poor (Day 14) | 2
  Q1: Missing (Day 14) | 18
  Q2: Very good (Day 14) | 16
  Q2: Good (Day 14) | 21
  Q2: Moderate (Day 14) | 19
  Q2: Poor (Day 14) | 3
  Q2: Very poor (Day 14) | 3
  Q2: Missing (Day 14) | 18
  Q3: Very good (Day 14) | 3
  Q3: Good (Day 14) | 8
  Q3: Moderate (Day 14) | 38
  Q3: Poor (Day 14) | 13
  Q3: Very poor (Day 14) | 0
  Q3: Missing (Day 14) | 18
  Q1: Very good (Day 28) | 3
  Q1: Good (Day 28) | 15
  Q1: Moderate (Day 28) | 21
  Q1: Poor (Day 28) | 7
  Q1: Very poor (Day 28) | 3
  Q1: Missing (Day 28) | 31
  Q2: Very good (Day 28) | 16
  Q2: Good (Day 28) | 16
  Q2: Moderate (Day 28) | 13
  Q2: Poor (Day 28) | 4
  Q2: Very poor (Day 28) | 0
  Q2: Missing (Day 28) | 31
  Q3: Very good (Day 28) | 3
  Q3: Good (Day 28) | 17
  Q3: Moderate (Day 28) | 21
  Q3: Poor (Day 28) | 8
  Q3: Very poor (Day 28) | 0
  Q3: Missing (Day 28) | 31
  Q1: Very good (Day 56) | 4
  Q1: Good (Day 56) | 18
  Q1: Moderate (Day 56) | 19
  Q1: Poor (Day 56) | 10
  Q1: Very poor (Day 56) | 1
  Q1: Missing (Day 56) | 28
  Q2: Very good (Day 56) | 14
  Q2: Good (Day 56) | 21
  Q2: Moderate (Day 56) | 9
  Q2: Poor (Day 56) | 4
  Q2: Very poor (Day 56) | 4
  Q2: Missing (Day 56) | 28
  Q3: Very good (Day 56) | 4
  Q3: Good (Day 56) | 16
  Q3: Moderate (Day 56) | 25
  Q3: Poor (Day 56) | 7
  Q3: Very poor (Day 56) | 0
  Q3: Missing (Day 56) | 28

ADVERSE EVENTS:
Time Frame: Baseline up to Day 56
Description: An adverse event is any untoward medical occurrence in a clinical study participant administered with study treatment. It can be any unfavorable and unintended sign/abnormal finding, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Arm/Group | Tramadol Hydrochloride/Acetaminophen
Serious Adverse Events (participants affected / at risk) | 2/80
Other Adverse Events (participants affected / at risk) | 49/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tramadol Hydrochloride/Acetaminophen (N=80)
Forearm fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tramadol Hydrochloride/Acetaminophen (N=80)
Palpitations (Cardiac disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Dry mouth (Gastrointestinal disorders) | 12
Flatulence (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 3
Chest pain (General disorders) | 2
Malaise (General disorders) | 1
Pain (General disorders) | 1
Dermatomyositis (Immune system disorders) | 2
Drug eruption (Immune system disorders) | 3
Nasopharyngitis (Infections and infestations) | 1
Gout (Metabolism and nutrition disorders) | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 14
Headache (Nervous system disorders) | 1
Vertigo (Nervous system disorders) | 4
Akathisia (Psychiatric disorders) | 1
Anorexia (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Decreased appetite (Psychiatric disorders) | 2
Sleep disorder (Psychiatric disorders) | 1
Somnolence (Psychiatric disorders) | 5
Dysuria (Renal and urinary disorders) | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Vascular disorders) | 1
Adenoviral upper respiratory (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less